CLINICAL TRIAL: NCT00534001
Title: A Phase II Study of the Effects of Extended Pre-Cessation Bupropion for Smoking Cessation
Brief Title: Bupropion in Helping Adults Stop Smoking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CDR0000565103; I 57805 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2015-08

CONDITIONS: Bladder Cancer; Cervical Cancer; Esophageal Cancer; Gastric Cancer; Head and Neck Cancer; Kidney Cancer; Leukemia; Liver Cancer; Lung Cancer; Pancreatic Cancer; Tobacco Use Disorder
Keywords: bladder cancer; cervical cancer; esophageal cancer; gastric cancer; renal cell carcinoma; adult primary liver cancer; non-small cell lung cancer; small cell lung cancer; pancreatic cancer; hypopharyngeal cancer; laryngeal cancer; lip and oral cavity cancer; nasopharyngeal cancer; oropharyngeal cancer; paranasal sinus and nasal cavity cancer; adult acute myeloid leukemia; tobacco use disorder
MeSH Terms: conditions — Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Leukemia; Liver Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Tobacco Use Disorder; Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Leukemia, Myeloid, Acute | interventions — Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (1-week run-in) (Experimental): Participants receive an oral placebo once or twice daily in weeks 1-3 followed by oral bupropion hydrochloride once or twice daily in week 4. Participants also undergo 90-minute behavioral group counseling sessions once in weeks 1, 2, and 4.
  Interventions: Drug: bupropion hydrochloride; Other: placebo
- Arm II (4-week run-in) (Experimental): Participants receive oral bupropion hydrochloride once or twice daily in weeks 1-4. Participants also undergo 90-minute behavioral group counseling sessions once in weeks 1, 2, and 4.
  Interventions: Drug: bupropion hydrochloride

INTERVENTIONS:
Drug: bupropion hydrochloride — Given orally
Other: placebo — Given orally
  Arms: Arm I (1-week run-in)

SUMMARY:
RATIONALE: Bupropion may help people stop smoking by decreasing the symptoms of nicotine withdrawal. Giving bupropion over a longer period of time may be effective in helping people stop smoking.

PURPOSE: This randomized phase II trial is studying how well bupropion works in helping adults stop smoking.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of conducting a full-scale clinical trial to evaluate whether extending the duration of pre-cessation bupropion hydrochloride enhances smoking cessation, as measured by 3-month prolonged abstinence rates, in adult smokers.

Secondary

* Assess baseline smoking and mood characteristics (nicotine dependence, smoking history, anxiety, and depression).
* Assess measures to address the hypothesized extinction mechanism (subjective effects of smoking, collection of cigarette butts for an assessment of nicotine and tar exposure, craving for smoking, and expectations for the consequences of smoking).
* Assess changes in affective state as measured by Withdrawal Symptoms Checklist and by Positive and Negative Affect Schedule (PANAS) questionnaire.
* Assess side effects, pill counts, and changes in daily smoking rate.
* Assess mental health, personality traits, interpersonal skills, demand simulation, impulsivity, motivation, and perceived stress using validated measures.

OUTLINE: Participants are stratified according to gender. Participants are randomized to 1 of 2 pre-cessation intervention arms.

* Arm I (1-week run-in): Participants receive an oral placebo once or twice daily in weeks 1-3 followed by oral bupropion hydrochloride once or twice daily in week 4. Participants also undergo 90-minute behavioral group counseling sessions once in weeks 1, 2, and 4.
* Arm II (4-week run-in): Participants receive oral bupropion hydrochloride once or twice daily in weeks 1-4. Participants also undergo 90-minute behavioral group counseling sessions once in weeks 1, 2, and 4.

In both arms, participants are asked to quit smoking (target quit date) in week 5. All participants then receive oral bupropion hydrochloride once or twice daily in weeks 5-11 and undergo 90-minute behavioral group counseling sessions once in weeks 5, 7, and 9.

Participants complete questionnaires to collect information on tobacco use history, health habits, depression, anxiety scales/symptoms, and sociodemographics at baseline. Participants also complete a series of validated questionnaires about smoking patterns, smoking satisfaction, mental health, personality traits, interpersonal skills, demand simulation, impulsivity, motivation, and perceived stress at baseline and then periodically during study. Participants undergo saliva sample collection at baseline and then periodically during study. Samples are analyzed for the presence of cotinine. Buccal cells are also collected at baseline for subsequent DNA analyses. Cigarette butts from the first cigarette of the day, including the quit day, are collected during group counseling sessions in weeks 1, 2, 4, and 5 and are assessed for a marker that indicates the amount of nicotine and tar consumed.

After finishing study treatment, participants are followed at 6 and 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Currently smokes ≥ 15 cigarettes per day for at least 1 year
* Motivated to quit smoking within the next 3 months

PATIENT CHARACTERISTICS:

* Willing to attend clinic visits
* Willing to refrain from nicotine replacement therapy (NRT) use during study participation
* Able to speak and read English fluently
* Has a home telephone and plans to reside in Western New York for the next year
* Not pregnant or nursing
* Negative pregnancy test
* Not planning a pregnancy
* Fertile patients must use effective contraception during and for 3 months after study participation
* No history of chronic renal or hepatic disease
* No history of head trauma or seizure
* No history of a seizure disorder, brain tumor, or CNS tumor
* No history of or currently diagnosed bulimia or anorexia nervosa
* No history of psychotic disorder
* No diabetes requiring oral hypoglycemics or insulin
* No excessive use of alcohol or alcoholism
* No current addiction to opiates, cocaine, or stimulants
* No poorly controlled hypertension (i.e., systolic blood pressure [BP] > 170 mm Hg and/or diastolic BP > 110 mm Hg)
* No allergy to bupropion hydrochloride
* No other surgical or medical condition that may significantly alter absorption, distribution, metabolism, or excretion of bupropion hydrochloride
* No history of noncompliance to medical regimens
* No other clinical contraindication
* No major depressive disorder

PRIOR CONCURRENT THERAPY:

* At least 14 days since prior and no concurrent monoamine oxidase inhibitor
* No recent discontinuation of a benzodiazepine
* No concurrent Hypericum perforatum (St. John's wort)
* No other concurrent drugs containing bupropion hydrochloride (e.g., Wellbutrin or Zyban)
* No concurrent antipsychotics, antidepressants, theophylline, systemic steroids, over-the-counter stimulants or anorectics, or levodopa
* No concurrent active treatment for cancer (e.g., chemotherapy or radiotherapy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Mahoney, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1-week Run In (Standard) | 4-week Run-in (Extended)
Started | 48 | 47
Completed | 43 | 43
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (1-week run-in) | Arm II (4-week run-in) | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (9.3) | 45.8 (10.1) | 46 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 50
  Male | 22 | 23 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Racial/Ethnic Minority | 5 | 4 | 9
  White/Not Hispanic | 43 | 43 | 86
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48 | 47 | 95
Cigarettes Smoked Per Day (CPD) [Mean (Standard Deviation); unit: CPD] | 22.0 (6.0) | 23.4 (7.9) | 23 (7)

OUTCOME MEASURES:

1. Primary Outcome: Prequit Change in Cigarettes Per Day
Description: Prequit Change in Cigarettes Per Day
Time Frame: 3-Week PreQuit Drug Manipulation Phase
Population: Excludes participants with missing data (2 in Arm 1, 3 in Arm 2)
Measure: Mean (Standard Error); unit: Cigarettes Per Day
Arm/Group | Arm I (1-week run-in) | Arm II (4-week run-in)
Number analyzed (Participants) | 46 | 46
Cigarettes Per Day | -2.6 (0.5) | -3.9 (0.6)

2. Secondary Outcome: Abstinence
Description: Bioverified 4-week continuous abstinence
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (1-week run-in) | Arm II (4-week run-in)
Number analyzed (Participants) | 48 | 47
Participants | 25 | 15

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Only participant-volunteered side effects were noted.
Arm/Group | Arm I (1-week run-in) | Arm II (4-week run-in)
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 48/48 | 47/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (1-week run-in) (N=48) | Arm II (4-week run-in) (N=47)
Any Non-Serious Adverse Event (General disorders) | 48 (48) | 47 (47) — Adverse events (not including serious) only tracked for clinical monitoring; all participants noted at least one adverse event during the 8-week period of monitoring.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No